CLINICAL TRIAL: NCT01529190
Title: Effect of Preoperative Pregabalin on Pain Intensity and Interleukin-6 Levels in Living Donor Kidney
Brief Title: Pregabalin on Interleukin-6 Levels in Living Donor Kidney
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Ellen de Queiroz Santiago, medical resident, principal investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pregabalin
Record Dates: First submitted 2011-10-03; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2011-12

CONDITIONS: Pain
Keywords: pregabalin; postoperative pain control; interleukin-6; acute pain
MeSH Terms: conditions — Pain; Acute Pain | interventions — Pregabalin; Pain Clinics; Interleukin-6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pregabalin 300mg (Active Comparator): Group 1 patients will receive a single dose of 300 mg pregabalin, 1 hour before the surgical incision; group 2 patients will receive a placebo dose. Pain intensity will be assessed with the numeric rating scale. The consumption of tramadol in 24 hours after surgery and the time for the first complementation dose will be registered. Blood samples will be collected by 6 hours and 24 hours after surgical incision, for IL-6 dosage, and maintained at -70 celsus degree
  Interventions: Drug: Pregabalin
- sugar pill (Placebo Comparator): group 2 will receive a placebo dose, 1 hour before tue surgical icnision
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Effect of Preoperative Pregabalin on Pain Intensity. 300mg of pregabalin before surgical incision
  Other Names: acute pain; interleukin-6
  Arms: pregabalin 300mg
Drug: Placebo — placebo
  Arms: sugar pill

SUMMARY:
Pregabalin, a ligand for alfa2delta subunits of voltage-gated calcium channels, has been shown to be an effective adjuvant therapy for acute postoperative pain, by inhibiting central sensitization. The IL-6, is detectable 60 minutes after surgical incision, persisting for until 10 days, with maximal plasmatic level in 4 and 6 hours. The objective of this study is evaluating the analgesic effect of pregabalin and its repercussion on serum levels of IL6.

DETAILED DESCRIPTION:
After approved by the Ethical Committee and signed informed consent, 40 patients aged from 18 until 60 years undergoing nephrectomy will be randomized in two groups. Group 1 patients will receive a single dose of 300 mg pregabalin, 1 hour before the surgical incision; group 2 patients will receive a placebo dose. Pain intensity will be assessed with the numeric rating scale. The consumption of tramadol in 24 hours after surgery and the time for the first complementation dose will be registered. Blood samples will be collected by 6 hours and 24 hours after surgical incision, for IL-6 dosage, and maintained at -70 celsus degree. The IL-6 dosages will be performed by the ELISA (enzyme-linked immunosorbent assay) method. The number of patients was calculated by Instat Graph® program. To detect difference in pain intensity of 3 between the groups by NRS, with 95% of power (estimated SD= 2.0), when the alpha level is set at 0.05, the sample should be of 20. Statistical analyses will be performed with parametric and nonparametric tests, considering the variety studied. The statistical program that will be utilized is Instat Graph®.

ELIGIBILITY:
Inclusion Criteria:

* living donor kidney

Exclusion Criteria:

* myocardial ischemia
* psychiatric disease
* absence of chronic pain
* absence of drugs dependency
* don´t use of opioid medication 1 week before surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Effect of preoperative pregabalin on pain intensity in living donor kidney | first 24 hours after surgery

SECONDARY OUTCOMES:
Effect of preoperative pregabalin on interleukin-6 levels in living donor kidney | first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Taylor CP. Mechanisms of analgesia by gabapentin and pregabalin--calcium channel alpha2-delta [Cavalpha2-delta] ligands. Pain. 2009 Mar;142(1-2):13-6. doi: 10.1016/j.pain.2008.11.019. Epub 2009 Jan 6. No abstract available. PMID 19128880
- [Background] Gray P, Kirby J, Smith MT, Cabot PJ, Williams B, Doecke J, Cramond T. Pregabalin in severe burn injury pain: a double-blind, randomised placebo-controlled trial. Pain. 2011 Jun;152(6):1279-1288. doi: 10.1016/j.pain.2011.01.055. Epub 2011 Mar 12. PMID 21398038
- [Background] Baidya DK, Agarwal A, Khanna P, Arora MK. Pregabalin in acute and chronic pain. J Anaesthesiol Clin Pharmacol. 2011 Jul;27(3):307-14. doi: 10.4103/0970-9185.83672. PMID 21897498